CLINICAL TRIAL: NCT02513797
Title: Left Atrial Appendage Ligation With the LARIAT™ Suture Delivery System as Adjunctive Therapy to Pulmonary Vein Isolation for Persistent or Longstanding Persistent Atrial Fibrillation
Brief Title: aMAZE Study: LAA Ligation Adjunctive to PVI for Persistent or Longstanding Persistent Atrial Fibrillation
Acronym: aMAZE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS-011; NCT02631915 (obsolete NCT alias)
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LARIAT + PVI Treatment Group (Experimental): Percutaneously isolate and ligate the Left Atrial Appendage (LAA) from the left atrium (LA) with the LARIAT System prior to planned pulmonary vein isolation (PVI) catheter ablation
  Interventions: Device: LARIAT + PVI; Device: Pulmonary Vein Isolation
- PVI Catheter Ablation Group (Active Comparator): Perform pulmonary vein isolation (PVI) catheter ablation procedure using a contact force sensing, irrigated radiofrequency catheter approved by FDA for the treatment of atrial fibrillation.
  Interventions: Device: Pulmonary Vein Isolation

INTERVENTIONS:
Device: LARIAT + PVI — Left Atrial Appendage ligation with the LARIAT System initially performed followed by adjunctive pulmonary vein isolation catheter ablation in staged procedures
  Other Names: Left Atrial Appendage ligation + Pulmonary Vein Isolation
  Arms: LARIAT + PVI Treatment Group
Device: Pulmonary Vein Isolation — Perform pulmonary vein isolation (PVI) catheter ablation procedure using a contact force sensing, irrigated radiofrequency catheter approved by FDA for the treatment of atrial fibrillation.

SUMMARY:
This study is a prospective, multicenter, randomized (2:1) controlled study to evaluate the safety and effectiveness of the LARIAT System to percutaneously isolate and ligate the Left Atrial Appendage from the left atrium as an adjunct to planned pulmonary vein isolation (PVI) catheter ablation in the treatment of subjects with symptomatic persistent or longstanding persistent atrial fibrillation.

This study will be conducted in two stages:

* Limited Early Stage (Stage 1): up to 250 subjects at up to 65 sites. (COMPLETED, transitioned to Stage 2)
* Pivotal Stage/ Phase III (Stage 2): up to 600 subjects at up to 65 sites. (COMPLETED) All subjects from both stages will be included in the primary analysis.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of symptomatic continuous persistent or longstanding persistent non-valvular atrial fibrillation
* Failed at least one Class I or III Antiarrythmic drug (AAD) and therefore, eligible and intended for standard of care catheter ablation;
* Life expectancy ≥ 1 year;
* Willing and able to return to and comply with scheduled follow-up visits and tests; and
* Willing and able to provide written informed consent

Exclusion Criteria:

* Prior procedure involving opening of the pericardium or entering the pericardial space (e.g., coronary artery bypass graft, heart transplantation, valve surgery) where adhesions are suspected;
* Any prior epicardial ablation or any type of left-sided atrial ablation procedure;
* LA diameter > 6 cm as measured by computerized tomography and confirmed by the imaging core laboratory;
* Documented embolic stroke, transient ischemic attach or suspected neurologic event within 3 months prior to the planned study intervention;
* Currently exhibits New York Heart Association Class IV heart failure symptoms;
* Documented history of right heart failure specifically when right ventricle exceeds the left ventricular size;
* Documented history of myocardial infarction (MI) within 3 months prior to the planned study intervention;
* Documented history of unstable angina within 3 months prior to the planned study intervention;
* Documented history of cardiogenic shock, hemodynamic instability or any medical condition in which intra-aortic balloon pump (IABP) therapy is clinically indicated within 3 months prior to the planned study intervention;
* Documented symptomatic carotid disease, defined as > 70% stenosis or > 50% stenosis with symptoms;
* Diagnosed active local or systemic infection, septicemia or fever of unknown origin at tme of baseline screening;
* Chronic renal insufficiency defined as eGFR < 30 mL/min/1.73m2 within 3 months prior to planned study intervention;
* End Stage Renal Disease (ESRD) or documented history of renal replacement / dialysis;
* Current documented history of clinically significant liver disease which predisposes the subject to significant bleeding risk (clinically defined by the treating physician);
* Any history of thoracic radiation with the exception of localized radiation treatment for breast cancer;
* Current documented use of long-term treatment with oral corticoid steroids, not including use of inhaled steroids for respiratory diseases;
* Active pericarditis;
* Active endocarditis;
* Any documented history or autoimmune disease associated with pericarditis;
* Evidence of Pectus Excavatum (documented and clinically defined by the treating physician);
* Untreated severe scoliosis (documented and clinically defined by treating physician);
* Documented Left Ventricular Ejection Fraction (LVEF) < 30% within 30 days prior to planned intervention;
* Documented presence of implanted congenital defect closure devices, (e.g., atrial septal defect, patent foramen ovale or ventricular septal defect device);
* Previously attempted occlusion of the left atrial appendage (by any surgical or percutaneous method);
* Inability, or unwillingness or contraindication to undergo TEE or CTA imaging or 24-hour Holter monitoring;
* Body Mass Index (BMI) > 40;
* Evidence of active Graves disease;
* Current untreated hypothyroidism;
* Any contraindication to suture, endovascular device, or other minimally invasive techniques including percutaneous, transseptal, and/or sub-xiphoid access;
* Subject is pregnant or plans / desires to get pregnant within next 12 months;
* Current enrollment in an investigation or study of an investigational device or investigational drug that would interfere with this study and the required follow up;
* Mental impairment or other psychiatric conditions which may not allow patient to understand the nature, significance and scope of the study;
* Any other criteria, medical illness or comorbidity which would make the subject unsuitable to participate in this study as determined by the clinical site Primary Investigator;

Additional Exclusion Criteria: Based on Screening / Pre-procedure Imaging

Subjects will also be excluded if they meet any of the following:

* Based on screening computed tomography angiography performed within 90 days prior to study intervention as confirmed by the core lab:

  * Left atrial appendage morphology: Superior-posterior oriented left atrial appendage (i.e. superior C shape), that has Left atrial appendage distal apex extending posterior to the ostium of the appendage.
  * Left atrial appendage positioned behind the pulmonary artery; or
  * All other left atrial morphology: Left atrial appendage LARIAT approach width > 50 mm.
* Based on a peri-procedural imaging (transesophageal echocardiography) at time of LARIAT or catheter ablation) and confirmed by institution's designated LARIAT echocardiographer:

  * Intracardiac thrombus; or
  * Significant mitral valve stenosis (i.e., mitral valve stenosis < 1.5cm2)

NOTE: It is anticipated that a majority of subjects enrolled in the aMAZE Trial will be elderly US Medicare beneficiaries. Therefore, the results from the aMAZE Trial are expected to be generalizable to the Medicare population.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Freedom from episodes of atrial fibrillation > 30 seconds at 12 months post index pulmonary vein isolation | 12 months following Pulmonary Vein Isolation catheter ablation procedure
  Measured by 24-hour Holter Monitoring

SECONDARY OUTCOMES:
Freedom from any atrial fibrillation/atrial tachycardia/atrial flutter recurrence defined as any episode > 30 seconds with or without AAD | Following the 90 day blanking period through 12 months post-index pulmonary vein isolation
  Measured by 24-hour Holter Monitoring
Composite endpoint of stroke of any cause and systemic embolism as adjudicated by the clinical events committee | 12 months following index pulmonary vein isolation

OTHER OUTCOMES:
LARIAT Technical Success | Immediately post-LARIAT ligation (acute) and at 12 months following index pulmonary vein isolation
  Successful placement of the LARIAT device pre-tied suture around the left atrial appendage to achieve left atrial appendage ligation defined as ≤1 ± 1mm diameter residual communication w/ left atrium, as assessed by transesophageal echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: David J Wilber, MD, Study Chair — Loyola University Department of Medicine; Dhanunjaya Lakkireddy, MD, Study Chair — Kansas City Cardiac Arrhythmia Research
Locations (53):
- United States (53):
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Scripps Clinic, La Jolla, California
  - University of California San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Stanford University, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - St. Vincent's HealthCare, Jacksonville, Florida
  - Piedmont Athens Regional Cardiology, Athens, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern University / Bluhm Cardiovascular Institute, Chicago, Illinois
  - Loyola University Center for Heart and Vascular Medicine, Maywood, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Community Hospital, Munster, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Kansas City Cardiac Arrhythmia Research, Overland Park, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Cardiovascular Institute of the South Clinical Research Corporation, Houma, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - UP Health System- Marquette, Marquette, Michigan
  - St. Luke's Hospital, Kansas City, Missouri
  - DaVita Medical Group, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - New York University Langone Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Ohio Health Research Institute, Columbus, Ohio
  - Southern Oregon Cardiology, Medford, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Bryn Mawr Medical Specialists Association / Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Austin Heart, Austin, Texas
  - Baylor - St. Luke's Medical Center, Houston, Texas
  - Houston Methodist, Houston, Texas
  - Baylor Plano Scott & White Research Institute Heart Hospital, Plano, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
  - Providence Sacred Heart Medical Center, Spokane, Washington

REFERENCES:
- [Background] Lee RJ, Lakkireddy D, Mittal S, Ellis C, Connor JT, Saville BR, Wilber D. Percutaneous alternative to the Maze procedure for the treatment of persistent or long-standing persistent atrial fibrillation (aMAZE trial): Rationale and design. Am Heart J. 2015 Dec;170(6):1184-94. doi: 10.1016/j.ahj.2015.09.019. Epub 2015 Oct 3. PMID 26678640
- [Derived] Lakkireddy DR, Wilber DJ, Mittal S, Tschopp D, Ellis CR, Rasekh A, Hounshell T, Evonich R, Chandhok S, Berger RD, Horton R, Hoskins MH, Calkins H, Yakubov SJ, Simons P, Saville BR, Lee RJ; aMAZE Investigators. Pulmonary Vein Isolation With or Without Left Atrial Appendage Ligation in Atrial Fibrillation: The aMAZE Randomized Clinical Trial. JAMA. 2024 Apr 2;331(13):1099-1108. doi: 10.1001/jama.2024.3026. PMID 38563835
- See also: aMAZE Trial website — http://amazetrial.com/